CLINICAL TRIAL: NCT02721277
Title: Compassionate Use of an Intravenous Fat Emulsion Comprised of Soy Oil, Medium Chain Triglycerides, Olive Oil, and Fish Oil for Neonates With Parenteral Nutrition Induced Liver Injury
Brief Title: SMOFlipid to Lessen the Severity of Neonatal Cholestasis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201600068
Record Dates: First submitted 2016-02-23; First posted 2016-03-29 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Cholestasis; Jaundice, Obstructive
Keywords: Parenteral nutrition, Total; Infant, newborn; Cholestasis; Enterocolitis, Necrotizing
MeSH Terms: conditions — Cholestasis; Jaundice, Obstructive; Hyperphagia; Enterocolitis, Necrotizing | interventions — SMOFlipid; Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SMOFlipid (Experimental): Subjects with cholestasis will receive 3 G/kg/day of intravenous SMOFlipid daily until parenteral nutrition (PN) is discontinued. In addition, the following monitoring for effects of SMOFlipid will be performed: total days of parenteral nutrition, maximum conjugated bilirubin, time to resolution of bilirubin, time to liver transplant, time to death, positive blood cultures, rates of increase in weight, length, and head circumference, time dependent changes in liver function tests, including triglycerides, and length of hospital stay.
  Interventions: Drug: SMOFlipid

INTERVENTIONS:
Drug: SMOFlipid — SMOFlipid contains a mixture of 4 different lipid sources: soybean oil which provides essential fatty acids, olive oil which is high in monounsaturated fatty acids that are less susceptible to lipid peroxidation than polyunsaturated fatty acids, medium-chain triglycerides which show a faster metabolic clearance than long-chain triglycerides, and fish oil which provides the supply of omega-3 fatty acids.
  Other Names: Parenteral nutrition (PN)

SUMMARY:
Parenteral nutrition (PN) provides intravenous nutritional supplementation for infants unable to absorb adequate enteral nutrients secondary to insufficient intestinal length or function. In early PN-associated cholestasis, the dose of traditional soy based lipid is limited to 1 g/kg/day which often limits the growth capacity of parenteral nutrition-dependent infants. Inadequate growth is directly related to poor neurological outcomes, failure to facilitate mechanical ventilation, and less growth of the neonate's already damaged intestine. Ultimately, these outcomes can lead to severe disability and death. To mitigate these deleterious effects and optimize growth, parenteral nutrition-dependent infants with cholestasis who are not adequately growing on 1 g/kg/day of soy-based lipid emulsion must have a greater intake of lipids to meet their needs for weight, length, and head circumference growth.

SMOFlipid contains a mixture of 4 different lipid sources: soybean oil which provides essential fatty acids, olive oil which is high in monounsaturated fatty acids that are less susceptible to lipid peroxidation than polyunsaturated fatty acids, medium-chain triglycerides which show a faster metabolic clearance than long-chain triglycerides, and fish oil which provides the supply of omega-3 fatty acids. The utility of Omegaven and soy-based lipid emulsion is limited as these are restricted to 1 g/kg/day in cholestatic infants. SMOFlipid is safe to be provided at the usual goal infusion amount of 3 g/kg/day. Because this product includes both omega-6 and omega-3 lipids, it provides the benefits of the omega-3s for the liver and provides more than enough omega-6s to meet essential fatty acid requirements. Its use in situations in which growth is inadequate in babies who must be restricted to 1 g/kg/day can be expected to improve their growth and likely markedly increase their chances of both a good neurological outcome and survival.

The aim of this research study is to determine if the unique formulation of SMOFLipid will cause less hepatic inflammation compared to soy only intralipids.

DETAILED DESCRIPTION:
The neonates who are being treated at the University of Florida Health Neonates Intensive Care Unit and are anticipated to need more than 21 days of intravenous nutrition will be considered as potential subjects. These subjects will receive the unique formulation of SMOFLipid

The following data will be collected from the subject's EMR by members of the research team:

* Lab values that evaluate liver function
* Growth parameters like head circumference, length, weight
* Medical/surgical history
* Time to resolution of bilirubin, time to liver transplant, time to death
* Length of hospital stay
* Rates of blood infections

Subjects will remain on SMOFlipid until weaned from PN.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 14 days old and less than 1 year of age.
* Greater than 1 kg.
* Mild cholestasis, defined as a conjugated bilirubin between 0.5-1.9 mg/dL
* Currently standard therapy with soy-based Intralipid
* Evidence of growth of weight, head circumference or length below our standards for post-menstrual age for at least 1 week.
* Be expected to require intravenous nutrition for at least an additional 21 days

Exclusion Criteria:

* Have a congenitally lethal condition.
* Have clinically severe bleeding or clinical liver failure not able to be managed with routine measures.
* Have evidence of a viral hepatitis or primary liver disease as the primary etiology of their cholestasis.
* Have other health problems such that survival is extremely unlikely even if the infant's cholestasis improves

Ages: 23 Weeks to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Neu, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SMOFlipid
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SMOFlipid
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Inflammation of the Liver Between the Groups
Description: Inflammation of the liver will be evaluated by comparing direct bilirubin values between the two groups.
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

2. Secondary Outcome: Measurement of Head Circumference for Growth Increase
Description: Growth increase will be measured by head circumference of participants.
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

3. Secondary Outcome: Measurement of Weight for Growth Increase
Description: Growth increase will be measured by weight of participants.
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

4. Secondary Outcome: Measurement of Length for Growth Increase
Description: Growth increase will be measured by length of participants.
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Subjects Requiring Surgery
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Concomitant Medications Received
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

7. Secondary Outcome: Length of IV Nutritional Therapy
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Subjects Receiving Formula Diet
Description: Enteral administration of formula will be noted
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Subjects Receiving Breast Milk Diet
Description: Enteral administration of breast milk will be noted
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Adverse Events Related to Treatment
Description: Laboratory values will be used to determine adverse events.
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

11. Secondary Outcome: Carbon Dioxide Total
Description: Laboratory value that determines acid-base balance
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

12. Secondary Outcome: Total Protein
Description: Laboratory value that evaluates liver function
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

13. Secondary Outcome: Albumin
Description: Laboratory value that evaluates liver function
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

14. Secondary Outcome: Aspartate Aminotransferase
Description: Laboratory value that evaluates liver function
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

15. Secondary Outcome: Alanine Aminotransferase
Description: Laboratory value that evaluates liver function
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

16. Secondary Outcome: Total Bilirubin
Description: Laboratory value that evaluates liver function
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

17. Secondary Outcome: Serum Glucose
Description: Laboratory values that evaluates glucose in the blood
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

18. Secondary Outcome: Alkaline Phosphatase
Description: Laboratory value that evaluates liver function
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

19. Secondary Outcome: Triglyceride
Description: Laboratory value that evaluates liver function and metabolism of fat
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Number of Days on Mechanical Ventilation Via Endotracheal Tube
Description: Length of therapy with mechanical ventilation
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

21. Other Pre Specified Outcome: Number of Days on Oxygen Via Continuous Positive Airway Pressure
Description: Length of therapy with nasal continuous positive airway pressure
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

22. Other Pre Specified Outcome: Number of Days on Oxygen Via Nasal Cannula
Description: Length of therapy with nasal cannula
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

23. Other Pre Specified Outcome: Number of Days With Central Venous Catheter
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

24. Other Pre Specified Outcome: Number of Blood Infections
Description: A review of the subject's medical record will determine the presence of bacterial, viral, or fungi colony-forming units (CFU) in the blood.
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

25. Other Pre Specified Outcome: Numbers of Blood Infection Obtained From a Venipuncture
Description: A review of the subject's medical record will determine the location from which positive blood cultures were obtained.
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

26. Other Pre Specified Outcome: Numbers of Blood Infection Obtained From a Central Venous Catheter
Description: A review of the subject's medical record will determine the location from which positive blood cultures were obtained.
Time Frame: 6 months
Population: Study was terminated due to insufficient enrollment
Arm/Group | SMOFlipid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: <1 year
Arm/Group | SMOFlipid
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes